CLINICAL TRIAL: NCT01426815
Title: Exploration of TNF-alpha Blockade With Golimumab in the Induction of Clinical Remission in Patients With Early Peripheral Spondyloarthritis (SpA) According to ASAS-criteria
Acronym: CRESPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Janssen Biologics B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/529
Record Dates: First submitted 2011-08-30; First posted 2011-08-31 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Peripheral Spondylarthritis
Keywords: Peripheral spondylarthritis according to ASAS- criteria
MeSH Terms: interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Golimumab 50mg (Simponi ®) (Experimental)
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Placebo — The prefilled syringe with placebo will be administrated subcutaneously every 4 weeks during a study period of 24 weeks.
  Arms: Placebo
Drug: Golimumab — The prefilled syringe with golimumab 50mg (Simponi ®) will be administrated subcutaneously every 4 weeks during a study period of 48 weeks.
  Arms: Golimumab 50mg (Simponi ®)

SUMMARY:
In this Investigator Initiated study, the investigators want to explore the potential of an induction therapy with Tumor Necrosis Factor (TNF)-blocking agents in a very early disease stage (less than 3 months of symptom duration) of patients with predominant peripheral spondyloarthritis (SpA), classified according to the new Assessment of SpondyloArthritis (ASAS)-criteria. The hypothesis would be that treatment with a TNF-blocker at this early ("immature") stage of the disease would result in a significant higher number of patients in clinical remission compared to placebo, and that - comparable to the early Rheumatoid Arthritis (RA) patients in the BeSt-study - long-term treatment would not be necessary to maintain this remission in a number of patients.

In this placebo-controlled, double blind, randomized study (with open-label phase, starting at week 24) sixty patients fulfilling the Assessment of SpondyloArthritis (ASAS) criteria of peripheral spondylarthritis will be enrolled. Patients will be randomized in a 2:1 ratio (2 golimumab :1 placebo). During the placebo-controlled phase, 50mg golimumab, or placebo will be administrated subcutaneously (SC) every 4 weeks through week 20. Subjects will be treated with open-label Golimumab 50 mg SC injections at weeks 24, 28, 32, 36, 40, 44, and 48. If patients are in 'clinical remission' (clinical remission is defined by the absence of arthritis, enthesitis and dactylitis clinically at two major consecutive visits. Visits are planned at week 12, week 24, week 36 and week 48) then the treatment will be stopped. In case of clinical relapse, patients will be treated with open-label golimumab 50 mg SC. Patients in sustained clinical remission will be observed to assess the possibility of maintaining drug-free remission. The study duration will be 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for study participation if all of the following criteria are met:

* Subject is ≥ 18 years of age
* Subjects must meet the new Assessment of SpondyloArthritis (ASAS) criteria for peripheral spondyloarthritis:

  o Subjects must have current arthritis (asymmetric or predominantly in the lower limbs) or current enthesitis (except for enthesitis only along the spine, sacroiliac joints and/or chest wall) or current dactylitis PLUS:
* At least 1 of the following Peripheral Spondyloarthritis (SpA) features:

  * Anterior uveitis confirmed by an ophthalmologist(past or present)
  * Crohn's disease or ulcerative colitis diagnosed by a gastroenterologist (past or present)
  * Evidence of preceding infection (acute diarrhea or non-gonococcal urethritis or cervicitis 1month before arthritis)
  * Psoriasis diagnosed by a dermatologist (past or present)
  * Human Leukocyte Antigen (HLA) B27 positivity
  * Sacroiliitis by imaging defined as bilateral grade 2-4 or unilateral grade 3-4 sacroiliitis on plain radiographs, according to the modified New York criteria or active sacroiliitis on Magnetic Resonance Imaging (MRI) according to the ASAS consensus definition (ref of addendum)
* Subjects must have had onset of peripheral SpA symptoms ≤ 3 months prior to the screening visit
* Subjects must have active disease at screening and baseline, defined by Patient Global Assessment of Disease Activity Visual Analog Scale (VAS) ≥ 40mm and Patient Global Assessment of Pain VAS ≥ 40mm at screening and baseline visits.
* In subjects with concurrent axial SpA symptoms, the peripheral SpA symptoms must be the predominant symptoms at study entry based on the Investigator's clinical judgment.
* Subject has a negative Purified Protein Derivative (PPD) test (or equivalent) and Chest radiography (posteroanterior (PA) and lateral view) at screening. If the subject has a positive PPD test (or equivalent), has had a past ulcerative reaction of PPD placement and/or a Chest radiography consistent with prior TB exposure, the subject must initiate, or have documented completions of a course of anti-Tuberculosis therapy.
* Patients must undergo screening for Hepatitis B Virus (HBV) (this includes testing for HBsAg (Hepatitis B surface Antigen), anti-HBs (Hepatitis B surface antibody) and anti-HBc total (Hepatitis B core antibody total).
* Women of childbearing potential or men capable of fathering children must be using adequate birth control measures during the study and for 6 months after receiving the last administration of study agent. Female patients of childbearing potential must test negative for pregnancy.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or is of childbearing potential and is practicing an approved method of birth control throughout the study and for 6 months after last dose of study drug.

Examples of approved methods of birth control include the following:

* Condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD)
* Oral, parenteral or intravaginal contraceptives for 90 days prior to study drug administration
* A vasectomized partner

  * Subject is judged to be in good health as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination, chest x-ray (CXR), and a 12-lead electrocardiogram (ECG) performed during screening.
  * Subjects must be able and willing to provide written informed consent and comply with the requirements of this study protocol.
  * Subjects must be able and willing to self-administer sc injections or have a qualified person available to administer subcutaneous injections.

Exclusion Criteria:

* Medical history of inflammatory arthritis of a different etiology other than peripheral spondyloarthritis (e.g. rheumatoid arthritis, systemic lupus erythematosus, gout, or any arthritis with onset prior to age 16 years such as Juvenile idiopathic arthritis (JIA)).
* Prior exposure to any biologic therapy with a potential therapeutic impact on SpA, including anti-TNF therapy.
* Treatment with any investigational drug of chemical or biological nature within a minimum of 30 days or 5 half lives (whichever is longer) of the drug prior to the Baseline Visit.
* Infection(s) requiring treatment with intravenous (iv) anti-infectives within 30 days prior to the Baseline visit or oral anti-infectives within 14 days prior to the Baseline Visit.
* Have a known hypersensitivity to human immunoglobulin proteins or other components of golimumab.
* History of Central Nervous System (CNS) demyelinating disease or neurologic symptoms suggestive of CNS demyelinating disease.
* History of listeriosis, histoplasmosis, chronic of active Hepatitis B infection, Hepatitis C infection, human immunodeficiency virus (HIV) infection, immunodeficiency syndrome, chronic recurring infections or active TB.
* Have a history of, or concurrent, chronic heart failure, including medically controlled, asymptomatic Congestive Heart Failure (CHF).
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix.
* Have received, or are expected to receive, any live virus or bacterial vaccination within 3 months prior to the first administration of study agent, during the trial, or within 6 months after the last administration of study agent.
* Positive pregnancy test at screening or baseline.
* Female subjects who are breast-feeding or considering becoming pregnant during the study.
* History of clinically significant drug or alcohol abuse in the last 12 months.
* Clinically significant abnormal screening laboratory results as evaluated by the Investigator.
* Positive rheumatoid factor (RF) or anti-cyclic citrullinated peptide (anti-CCP) antibody at screening if the titers are crossing 3 times the upper limit of the normal
* Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.
* Subject with diagnosis and current symptoms of fibromyalgia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03-13 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Clinical remission | At 24 weeks
  The primary endpoint of the study is the induction of clinical remission (complete resolution of synovitis/dactylitis/enthesitis which was present at baseline) and prevention of newly developing peripheral and/or axial spondylarthritis signs). The primary analysis will be a comparison at 24 weeks of the percentage of patients in clinical remission in the group treated with the Tumor Necrosis Factor (TNF)-blocking agent versus placebo.

SECONDARY OUTCOMES:
The improvement in the tender and swollen joint count | At week 24.
  The key secondary endpoint will be the changes in the tender and swollen joint count (76/78 joint count)at 6 months (week 24) in comparison with baseline.
The improvement in dactylitis with obtaining a circumference measurement and clinical picture. | At week 24.
  The key secondary endpoint will be the changes in dactylitis at 6 months (week 24) in comparison with baseline.
The improvement in enthesitis, using the different scoring systems with inclusion of all relevant entheses. | At 24 weeks.
  The key secondary endpoint will be the changes in enthesitis at 6 months (week 24) in comparison with baseline.
The improvement in global measurements of disease activity. | At 24 weeks.
  The improvement in global measurements of disease activity: patient global assessment of disease activity, patient pain assessment (peripheral and axial pain), physician global assessment of disease activity, ...)
The exploration of the utility of conventional ankylosing spondylitis measurements such as BASDAI, BASFI, BASMI | At week 24.
  The key secundairy endpoints will be changes in global measurements of disease activity and conventional ankylosing spondylitis measurements (Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI),Bath Ankylosing Spondylitis Metrology Index (BASMI)) at 6 months (week 24) in comparison with baseline.
The exploration of the safety of (Tumor Necrosis Factor)TNF-α blockade in patients with early peripheral spondyloarthritis. | At 24 weeks.
  The improvement in global measurements of disease activity: patient global assessment of disease activity, patient pain assessment (peripheral and axial pain), physician global assessment of disease activity, ...)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Vandenbosch, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Krabbe S, Renson T, Jans L, Elewaut D, Van den Bosch F, Carron P, Ostergaard M. Performance of an MRI scoring system for inflammation of joints and entheses in peripheral SpA: post-hoc analysis of the CRESPA trial. Rheumatology (Oxford). 2023 Jun 1;62(6):2130-2138. doi: 10.1093/rheumatology/keac567. PMID 36200875
- [Derived] Carron P, De Craemer AS, Renson T, Colman R, Elewaut D, Van den Bosch F. TNFi-induced sustained clinical remission in peripheral spondyloarthritis patients cannot be maintained with a step-down strategy based on methotrexate. Rheumatology (Oxford). 2021 Oct 2;60(10):4880-4883. doi: 10.1093/rheumatology/keab056. PMID 33471112
- [Derived] Carron P, Varkas G, Renson T, Colman R, Elewaut D, Van den Bosch F. High Rate of Drug-Free Remission After Induction Therapy With Golimumab in Early Peripheral Spondyloarthritis. Arthritis Rheumatol. 2018 Nov;70(11):1769-1777. doi: 10.1002/art.40573. PMID 29806090
- [Derived] Carron P, Varkas G, Cypers H, Van Praet L, Elewaut D, Van den Bosch F; CRESPA investigator group. Anti-TNF-induced remission in very early peripheral spondyloarthritis: the CRESPA study. Ann Rheum Dis. 2017 Aug;76(8):1389-1395. doi: 10.1136/annrheumdis-2016-210775. Epub 2017 Feb 17. PMID 28213565
- See also: Related Info — http://www.uzgent.be